CLINICAL TRIAL: NCT00879411
Title: 24h BP Under Micardis in Daily Practice
Brief Title: Investigating the Effect of Telmisartan (Micardis®) on the Average 24h Blood Pressure of Therapy-naive and Therapy-experienced Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.582
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- arterial hypertension
  Interventions: Drug: Micardis

INTERVENTIONS:
Drug: Micardis

SUMMARY:
Practical experience report (PER) investigating the effect of Micardis® on the average 24h blood pressure of therapy-naive and therapy-experienced patients

ELIGIBILITY:
Inclusion criteria:

1. Patients who have recently been diagnosed with hypertension
2. Patients whose current blood pressure treatment are inadequate and needs to be revised are suitable for inclusion.

Exclusion criteria:

None (according to investigator)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telmisartan, Hydrochlorothiazide
Started | 701
Completed | 539
Not Completed | 162
Not completed — lost to follow-up (non-AE) | 162

BASELINE CHARACTERISTICS:
Arm/Group | Telmisartan, Hydrochlorothiazide
Number analyzed (Participants) | 701
Age, Continuous [Mean (Standard Deviation); unit: Year] | 60.5 (12.8)
Gender [Number; unit: participants] — 20 subjects did not indicate any specific gender
  participants
    Female | 324
    Male | 357
Baseline Diastolic Blood Pressure (DBP) values (ABPM) [Mean (Standard Deviation); unit: mm Hg] | 82 (9.6)
Baseline Systolic Blood Pressure (SBP) values (ABPM) [Mean (Standard Deviation); unit: mm Hg] | 136 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (Change of Systolic Blood Pressure)
Description: Change from baseline in 24h systolic blood pressure (BP) at week 8
Time Frame: baseline to 8 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Telmisartan, Hydrochlorothiazide
Number analyzed (Participants) | 537
mm Hg | 8.6 (17.8)

2. Primary Outcome: Efficacy (Change of Diastolic Blood Pressure)
Description: Change from baseline in 24h diastolic blood pressure (BP) at week 8
Time Frame: baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Telmisartan, Hydrochlorothiazide
Number analyzed (Participants) | 537
mm Hg | 4.7 (12.7)

3. Secondary Outcome: Overall Tolerability Scale
Description: Safety and tolerability of Micardis® in the treatment of patients with hypertension over 8 weeks, using 10 point Likert scale with worst score=1, best score=10
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telmisartan, Hydrochlorothiazide
Number analyzed (Participants) | 537
units on a scale | 9.2 (1.5)

ADVERSE EVENTS:
Time Frame: 56 Days
Arm/Group | Telmisartan, Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 0/701
Other Adverse Events (participants affected / at risk) | 0/701

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.